CLINICAL TRIAL: NCT00570180
Title: An Open-label Phase II Study of the Efficacy of Combination Bortezomib-containing Regimens in the Treatment of Newly Diagnosed Patients With t (4; 14) Positive Multiple Myeloma
Brief Title: Combination Bortezomib-containing Regimens in Newly Diagnosed Patients With t (4; 14) Positive Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Ortho Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-MMY-2016; t4;14 trial PMH (Other: Sponsor)
Record Dates: First submitted 2007-12-06; First posted 2007-12-10 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Please see intervention description for Bortezomib (Velcade)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — 21 day-cycle Induction therapy:bortezomib 1.3 mg/m2 (I.V. Days 1, 4, 8, and 11), then 10-day rest period. DOXIL 30 mg/m2 given after bortezomib (I.V. infusion Day 4 of each cycle). Dexamethasone 40 mg PO on days 1-4,8-11 and 15-18 during the first cycle. Subsequent 3 cycles, dexamethasone 40 mg PO given on days 1-4 and 11-14. Patients who don't progress may undergo elective stem cell mobilization, stem cell collection and cryopreservation. Patients will then receive post-induction therapy 1.5 mg/m2 bortezomib days 1, 8, and 15 I.V. + cyclophosphamide 300 mg/m2 PO weekly + prednisone 100 mg PO on alternate days for 8 monthly 28 day cycles.Maintenance therapy with weekly 40 mg dexamethasone (days 1, 8, 15 and 22) every month until disease progression occurs.
  Other Names: Velcade

SUMMARY:
Given the disappointing results with routine ASCT in t(4;14) patients, we propose this open label phase II study of bortezomib along with dexamethasone and pegylated liposomal doxorubicin (Doxil/Caelyx), referred to as the DBd regimen, for 4 cycles, followed by post-induction therapy with cyclophosphamide + bortezomib + prednisone (referred to as the CyBorP regimen) for 8 cycles. Since patients with t(4;14) remain at high risk for relapse, maintenance therapy with dexamethasone weekly will be given until disease progression.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS A. TITLE: An Open-Label Phase II Study of the Efficacy of Combination Bortezomib-containing Regimens in the Treatment of newly diagnosed patients with t (4;14) positive Multiple Myeloma.

B. RATIONALE: Between 15 and 20% of myeloma patients exhibit a t(4;14), which results in translocation of the receptor tyrosine kinase (TK) fibroblast growth factor receptor 3 (FGFR3) from chromosome 4 to the Immunoglobulin H (IgH) locus. The presence of a t(4;14) appears to confer an extremely poor prognosis. Patients with this abnormality do not experience prolonged remissions after a single autologous stem cell transplant (ASCT) using high-dose melphalan, and the optimal therapy of this group has not yet been defined. Specifically, data from Princess Margaret Hospital and the Mayo Clinic both indicate that the median progression-free survival (PFS) is only about 8 months and overall survival 18-22 months after ASCT. Unpublished data from the French Francophone Myeloma Intergroup (IFM) studies suggest that tandem transplants may improve these results modestly, but the outcome is still inferior compared with other cytogenetic subgroups.

Initial unpublished observations suggested that t(4;14) patients with relapsed/refractory disease were uniquely sensitive to the new agent bortezomib. More recent information in larger numbers of patients indicates that responses to single agent bortezomib are seen in up to 50-65% of t(4;14) patients; the duration of response is similar to that seen in other subsets, i.e. in the range of 5-7 months. Combinations of bortezomib with agents such as doxorubicin, pegylated liposomal doxorubicin, thalidomide, cyclophosphamide, melphalan, thalidomide and corticosteroids have been evaluated in a number of clinical studies in recurrent myeloma, and the response rates (RR) appear to be improved compared to single agent bortezomib, and toxicity has been acceptable.

In newly diagnosed myeloma patients, combinations such as vincristine, doxorubicin, dexamethasone (VAD) and thalidomide + dexamethasone are often utilized before ASCT. A study by Hussein et al. substituted pegylated liposomal doxorubicin for the conventional formulation of doxorubicin and noted a similar response rate with less grade 3/4 neutropenia, alopecia and sepsis; in addition, patients do not necessarily require a central venous catheter. More recently, Cavenagh et al. has reported remarkable activity with the so-called PAD regimen of bortezomib, doxorubicin and dexamethasone, with a combined Complete Remission (CR) + Partial Response (PR) rate of 67% following 1 cycle, and 93% after 4 cycles, with no impairment of the ability to collect blood stem cells for ASCT. Preliminary data from an ongoing Canadian phase II study of Doxil/Caelyx + Bortezomib + Dexamethasone (DBd), in which pegylated liposomal doxorubin, bortezomib and dexamethasone are combined, has produced encouraging results to date with minimal toxicity. In that study, DBd therapy was given for 4 cycles before ASCT independently of cytogenetic classification.

Given the disappointing results with routine ASCT in t(4;14) patients, we propose this open label phase II study of bortezomib along with dexamethasone and pegylated liposomal doxorubicin (Doxil/Caelyx), referred to as the DBd regimen, for 4 cycles, followed by post-induction therapy with cyclophosphamide + bortezomib + prednisone (referred to as the CyBorP regimen) for 8 cycles. Since patients with t(4;14) remain at high risk for relapse, maintenance therapy with dexamethasone weekly will be given until disease progression. This approach will test the hypothesis that bortezomib-based therapy can improve the outcome of newly diagnosed t(4;14) multiple myeloma patients.

C. OBJECTIVES OF THE STUDY: To evaluate the efficacy of the DBd regimen given as induction therapy, followed by post-induction therapy with CyBorP and maintenance therapy with dexamethasone in t(4;14) positive multiple myeloma (MM) patients.

Primary Objectives

* To determine the time to progression (TTP) with this treatment regimen. Secondary Endpoints
* To determine the objective response rate following DBd induction therapy
* To determine the duration of response following DBd induction therapy
* To determine the objective response rate following CyBorP post-induction therapy
* To determine the duration of response following CyBorP post-induction therapy
* To determine PFS
* To determine overall survival
* To determine the safety profile of this regimen
* To examine the ability of bortezomib based regimens to repress FGFR3 signaling

D. STUDY DESIGN: This is an open-label, Phase II study of induction therapy with bortezomib, pegylated liposomal doxorubicin (Doxil/Caelyx) and dexamethasone as initial therapy in patients with t(4;14). Each 21 day-cycle consists of bortezomib 1.3 mg/m2 (given as an I.V. bolus on Days 1, 4, 8, and 11) followed by a 10-day rest period (Days 12 to 21). DOXIL/CAELYX 30 mg/m2 will be given after bortezomib as at least a 1-hour I.V. infusion on Day 4 of each 21-day cycle. Dexamethasone 40 mg PO will be given on days 1-4, days 8-11 and days 15-18 during the first cycle. For the subsequent 3 cycles, dexamethasone 40 mg PO will be given on days 1-4 and days 11-14. Patients who do not experience disease progression may undergo elective, as per the attending physician's discretion, stem cell mobilization followed by stem cell collection and cryopreservation. Patients will then receive post-induction therapy with cyclophosphamide + bortezomib + prednisone (1.5 mg/m2 bortezomib on days 1, 8, and 15 I.V. + cyclophosphamide 300 mg/m2 PO weekly + prednisone 100 mg PO on alternate days) for 8 monthly 28 day cycles, followed by maintenance therapy with 40 mg of dexamethasone weekly per month until disease progression occurs.

E. PATIENT CHARACTERISTICS: Untreated multiple myeloma patients who are t(4;14) positive by fluorescence in situ hybridization (FISH) will be considered for the study. Exclusion criteria include inadequate liver function aspartate aminotransferase (AST} and alanine aminotransferase (ALT) > 2.5 times the upper limit of normal), thrombocytopenia (platelets < 50 X 109/L), neutropenia (absolute neutrophil count < 1.0 x 109/L), pregnant or lactating women, and women of childbearing potential (WCBP) who are not using adequate contraception and Left Ventricular Ejection Fraction (LVEF) below the institutional Lower Limit Normal (LLN) or less than 40%; whichever value is higher. A patient may have received up to 4 months of other anti myeloma therapy, as part of the induction therapy, prior enrollment and still be considered eligible to participate in the study, as long as the patient's multiple myeloma has not progressed in the current regimen and the other eligibility criteria are met.

F. STATISTICAL PLAN: The TTP from initiation of chemotherapy in patients treated with ASCT for this subset is approximately 12 months. An increase in TTP from 12 to 21 months would be of clinical significance. Using an 80% power to detect this time difference in a two-sided comparison patient, a sample size of 36 evaluable patients is required. This calculation assumes that each patient will be evaluated at a fixed time of 24 months. Assuming a 20% drop-out rate, a total sample size of 45 patients will be required.

G. STUDY DESIGN: It is assumed that the new regimen will not be of further interest in t(4;14) positive myeloma patients if the TTP from the time of starting induction therapy is less than 21 months. Each patient will be followed every month until disease progression and then after every 6 moths up to 5 years for survival. An interim analysis will also be performed after 12 patients have completed the post-induction therapy with cyclophosphamide + bortezomib + prednisone (CyBorP).

H. PATIENT ACCRUAL AND STUDY DURATION: Patients with t(4;14) represents only 15% of all myeloma patients, as such, accrual will be highly dependant on number of participating centers. It is estimated that approximately 350 newly-diagnosed patients will require cytogenetic screening in order to meet the accrual target. Accrual is expected to be complete within 48 months. Additional time is required, of course, to allow the response data to mature. All patients registered in the study will be accounted for (screen failures + enrolled patients). The number of patients who are not evaluable, who died or withdrew before treatment began will be specified. The distribution of follow-up times will be described and the number of patients lost to follow-up will be monitored.

I. EFFICACY PARAMETERS: Beginning in cycle 1, the response to treatment will be determined during each cycle using the International Myeloma Working Group uniform response criteria for multiple myeloma as outlined in Section 11.0. Responses will be assessed by monoclonal protein, monoclonal paraprotein (M protein) quantification from serum and a 24-hour urine collection (including immunofixation, if needed), bone marrow plasma cells, assessment of lytic lesions, and soft tissue plasmacytomas. For patients with light chain disease or non-secretory myeloma, a serum sample for Free Lite chain testing will be obtained and the results will be compared to the levels reported quantified in the urine.

J. REGISTRATION: Patients will be registered by completing the eligibility and enrollment checklist and forwarding it by fax to the Multiple Myeloma Research Coordinator at Princess Margaret Hospital at 416-946-4419, between the hours of 9 am and 4 pm Eastern Standard Time, up to 5 business days prior commencement of cycle 1 day 1. The research coordinator should also be contacted by phone at 416 946-4627. The checklist will be verified and a patient number will be assigned for eligible patients.

K. SAMPLE PROCESSING: Centralized screening will be employed at Princess Margaret Hospital. Following informed consent site should send two fresh heparinized (green top tube) marrow samples (5cc per tube or best available) by overnight courier (see Appendix VI for shipping and notification instructions) for t4;14 screening test. Tri-color fluorescence in situ hybridization (FISH) for t(4;14) will be performed and reported back to referring site within 5-7 working days.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with MM based on criteria from the International Myeloma Working Group (IMWG)
* Patients who have 'measurable' disease
* Age 18 years at the time of signing Informed Consent
* A patient may have received up to 4 months of other anti myeloma therapy, as part of the induction therapy, prior enrollment and still be considered eligible to participate in the study, as long as the patient's multiple myeloma has not progressed on the current regimen and the other eligibility criteria are met.
* Patient is t(4;14) positive on screening assay.

Exclusion Criteria:

* Concomitant therapy medications that include corticosteroids (> 10 mg per day of prednisone or equivalent) or other therapy that is or may be active against myeloma prior to day 1 (with the exception of radiation therapy or induction therapy as described under the above inclusion criteria section
* Peripheral neuropathy of Grade 2 or greater.
* Patients with evidence of mucosal or internal bleeding and/or refractoriness to platelet transfusions (i.e., unable to maintain a platelet count 50 x 109 /L).
* Patients with an absolute neutrophil count (ANC) < 1.0 x 109/L. Treatment to raise the ANC, such as granulocyte colony-stimulating factor (G-CSF) or granulocyte-macrophage colony-stimulating factor (GM-CSF) is not allowed within 14 days of study entry.
* Patients with hemoglobin < 80 g/L despite transfusion.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-08-25 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-15 (Actual)

PRIMARY OUTCOMES:
To determine the time to progression (TTP) with this treatment regimen | Patients were followed monthly until disease progression and subsequently every six months for up to five years to assess OS.
  Measured from the date of enrollment to the date of disease progression. Otherwise, censored at the time of last disease assessment. Responses were assessed using the International Myeloma Working Group criteria, involving a modified version of the European Group for Blood and Marrow Transplantation (EBMT) criteria, where the category of stringent complete response (sCR) was included for patients with normalization of the free light chain ratio.10,11 Bone marrow aspirate and biopsy were obtained routinely after induction therapy to confirm CR or sCR. Serum free light chain assay and serum and/or urine electrophoresis were performed monthly; immunofixation was performed when confirmation of very good partial response (VGPR), CR, or sCR was necessary.

SECONDARY OUTCOMES:
To determine the objective response rate/duration following DBd induction and Cybor P post induction therapy | Patients were followed monthly until disease progression
  Objective response after completing induction therapy and until disease progression.
To determine PFS | 5 years
  PFS was measured from the date of enrollment to the date of disease progression or death from any cause, otherwise censored at the time of last disease assessment.
To determine overall survival | 5 years
  Patients were followed monthly until disease progression and subsequently every six months for up to five years to assess OS.
To determine the safety profile of this regimen | 5 years
  Safety analyses focused on hematological and non-hematological adverse events of all grades. Toxicity was graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE version 3.0)

CONTACTS AND LOCATIONS:
Overall Officials: Donna E. Reece, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (7):
- Canada (7):
  - Cross Cancer Institute 11560 University Ave, Edmonton, Alberta
  - CancerCare Manitoba 675 McDermot Ave., Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre., Halifax, Nova Scotia
  - London Regional Cancer Program 790 Commissioners Road East, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Saskatoon Cancer Centre 20 Campus Drive, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
Un-identified data will be submitted to the DSMB for review. Sites will be provided with the DSMB letter after a meeting has been held to review data.